CLINICAL TRIAL: NCT03303209
Title: Patient-Centered Opioid Tapering in Outpatients With Chronic Pain and Long-Term Opioid Use
Brief Title: Patient-Centered Opioid Tapering Study
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Beth Darnall, Clinical Professor, Stanford University
Other Study IDs: 37179
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use; Chronic Pain
Keywords: opioid; opioids; taper; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient-centered opioid tapering protocol — All patients who entered the study agreed to partner with their pain physician on a patient-centered opioid tapering program. The research component of the study was to observe patient response (in terms of change in MEDD and pain intensity) at month 4.

SUMMARY:
This is an observational study of a voluntary opioid tapering protocol conducted in community outpatients taking long term prescription opioids for chronic pain. Patients who would otherwise continue with their existing opioid prescriptions were encouraged to participate in a voluntary opioid taper program. Interested patients were identified by their pain physician, Dr. Richard Stieg, and then completed an online informed consent document and baseline self-report assessments including types and doses of opioid medications as well as demographic and psychosocial measures, clinical and pain characteristics. Patients were either given or mailed a free copy of a patient book The Opioid-Free Pain Relief Kit, or Less Pain, Fewer Pills: Avoid the dangers of prescription opioids and gain control over chronic pain. Over the following weeks and up to 4 months, Dr. Stieg implemented a slow, individually tailored opioid taper in all patient participants. Follow-up online self-report surveys were completed at 4 months post enrollment. Opioid dose data were confirmed via medical chart review, and doses were converted to a standardized morphine equivalent daily dose (MEDD). Main outcome was change in opioid dose baseline to 4 months. Secondary outcome was change in pain intensity (numeric rating scale, 0-10) baseline to 4 months.

DETAILED DESCRIPTION:
Background: Background: An estimated 11 million Americans were prescribed long term opioids in 2014-up to 4 percent of the entire U.S. adult population. Patients with chronic pain taking long term opioids are at higher risk for multiple health problems including more severe pain and addiction, and death from accidental overdose. Opioid related overdoses are now a leading cause of death in the U.S. Multiple national agencies have called for reduced opioid prescriptions.

Lower doses of opioids are safer for patients. Patients who take very high dose opioids for chronic pain (>200 morphine equivalent daily dose; MEDD) are at 3-fold increased risk for accidental overdose death compared to those on low doses (1). However, the primary patient concern about reducing opioids is fear of having increased pain. Indeed, evidence is lacking for how to help real-world patients with chronic pain reduce opioid use while controlling their pain.

Inpatient studies suggest that pain improves with intensive pain rehabilitation and opioid cessation (2). interdisciplinary chronic pain rehabilitation combined with opioid cessation in veterans has been associated with improved indices of psychological and physical function, as well as significantly reduced pain in those who stop opioids during the program (3). However, inpatient and intensive opioid reduction programs are costly and unavailable to most patients. Recently, researchers conducted an outpatient randomized controlled trial comparing an outpatient opioid tapering program to usual care (4). The tapering program consisted of psychiatric consultation, opioid dose tapering, and 18 weekly meetings with a physician assistant to explore motivation for tapering and learn pain self-management skills.

No studies exist to inform best practice on opioid reduction in primary care or outpatient pain clinics. There is a critical gap in knowledge on how to help community-based (primary care and pain clinic) outpatients with chronic pain actively reduce opioids while controlling pain. This project was intended to inform real-world patient care to specifically help patients with chronic pain taking long term moderate-, high-, and super high-dose opioids reduce their daily use and associated risks. The goal is to understand whether a simple, patient-centered opioid taper conducted with limited resources and no interdisciplinary supportive treatments (e.g., psychology services, physical therapy) could effectively reduce opioid dose without increasing pain.

Methods

Study Design: A prospective observational study of a voluntary patient-centered opioid tapering program. The study was conducted in compliance with the Stanford University's Internal Review Board.

Participants: Adult patients with chronic pain prescribed opioids from a private practice pain clinic in Colorado were invited by their prescribing physician to participate in a voluntary opioid tapering program. Patients who expressed interest were called and invited into the study (note that the study, which involved collecting patient data, is distinct from the taper program. Patients could taper their opioids without agreeing to be studied). Inclusion criteria included adults over the age of 18 years, medically diagnosed chronic pain for at least 6 months, interest in participating in patient-centered opioid tapering, intact cognitive function, an absence of frank psychological disorder, able to speak/read English, able to complete online forms, and not being enrolled in a treatment program for substance use disorder.

Procedure

Patients from a private clinic with chronic pain using daily opioid medications were invited to participate in a voluntary opioid taper program by their physician. Those who agreed to participated were enrolled in the weaning program (taper program) with the physician. After patients provided informed consent, enrolled patients completed a series of online questionnaires that collect data on demographics, psychosocial factors, and physical, emotional, and cognitive function, and opioid medications (type and dose) at baseline and at 4-month follow-up. The opioid taper program was not regulated by the study protocol. It was supervised by the physician, and individually tailored to meet the patient's specific clinical needs. The goal was to reduce opioid consumption at a comfortable pace (individually determined) and target cessation at 4 months from the time they enter the weaning program.

Data Collected:

Demographics included age and gender. Clinical variables included opioid medications, length of time on opioids, pain diagnoses, pain intensity, and marijuana use (yes/no). Opioids were converted to a Morphine Equivalent Daily Dose (MEDD) using standard procedures. MEDDs were calculated for baseline and for the 4 month follow-up time point.

Current Medications Pain Catastrophizing Scale PROMIS Global Health Scale PROMIS Fatigue Scale PROMIS Pain Interference Scale PROMIS Physical Function Scale PROMIS Emotional Distress-Anxiety Scale PROMIS Depression Scale PROMIS Sleep Disturbance Scale PROMIS Sleep Interference PROMIS Pain Behavior Scale PROMIS Social Isolation PROMIS Sleep Related Impairment Scale PROMIS Cognitive Function Scale PROMIS Pain Intensity PROMIS Applied Cog Abilities Marijuana use (yes/no)

Analytic Plan:

Descriptive statistics will include means, medians, ranges, frequencies and percentiles for study variables.

For continuous variables: Welch Two Sample, two-sided t-test without assumption of equal variance will be used.

Polychotomous variables: Pearson's Chi-squared test with Yates' continuity correction. For cells with small numbers, P value will be simulated with 2000 replications.

PRIMARY OUTCOME:

Assuming the primary outcome MEDD will not be normally distributed, Kruskal-Wallis rank sum test will be used to compare MEDD at baseline and 16 weeks.

Pain intensity, our secondary outcome will be assessed similarly.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18
* Chronic pain
* Chronic daily opioids
* Wish to reduce opioid dose

Exclusion Criteria:

* Not able to communicate in English
* Not able to complete electronic questionnaires
* No major cognitive impairment
* Not actively engaged in treatment for substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain receiving treatment in a community chronic pain clinic who were also taking long term prescription opioids were invited by their prescribing physician to participate in patient-centered, voluntary opioid tapering.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Change in Morphine Equivalent Daily Dose (MEDD) from baseline to 4 months. | 4 months
  Pre-post MEDD change was calculated

SECONDARY OUTCOMES:
Change in Pain Intensity from baseline to 4 months | 4 months
  Pre-post changes in pain intensity (using the 0-10 numeric rating scale) were calculated

CONTACTS AND LOCATIONS:
Overall Officials: Beth Darnall, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No
We have no plan in place; however data may be shared upon request.

REFERENCES:
- [Background] Gomes T, Mamdani MM, Dhalla IA, Paterson JM, Juurlink DN. Opioid dose and drug-related mortality in patients with nonmalignant pain. Arch Intern Med. 2011 Apr 11;171(7):686-91. doi: 10.1001/archinternmed.2011.117. PMID 21482846
- [Background] Crisostomo RA, Schmidt JE, Hooten WM, Kerkvliet JL, Townsend CO, Bruce BK. Withdrawal of analgesic medication for chronic low-back pain patients: improvement in outcomes of multidisciplinary rehabilitation regardless of surgical history. Am J Phys Med Rehabil. 2008 Jul;87(7):527-36. doi: 10.1097/PHM.0b013e31817c124f. PMID 18574345
- [Background] Murphy JL, Clark ME, Banou E. Opioid cessation and multidimensional outcomes after interdisciplinary chronic pain treatment. Clin J Pain. 2013 Feb;29(2):109-17. doi: 10.1097/AJP.0b013e3182579935. PMID 22751033
- [Background] Sullivan MD, Turner JA, DiLodovico C, D'Appollonio A, Stephens K, Chan YF. Prescription Opioid Taper Support for Outpatients With Chronic Pain: A Randomized Controlled Trial. J Pain. 2017 Mar;18(3):308-318. doi: 10.1016/j.jpain.2016.11.003. Epub 2016 Nov 28. PMID 27908840